CLINICAL TRIAL: NCT05595096
Title: Comparison of Thoracic Paravertebral Nerve Block Combined Laryngeal Mask Airway With Preservation of Spontaneous Breathing Versus General Anesthesia Using Double-lumen Endobronchial Intubation in Patients Undergoing Thoracoscopic Surgery:
Brief Title: Preservation of Spontaneous Breathing in Patients Undergoing Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhenjiang First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y2021017
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Thoracoscopic Surgery
Keywords: Spontaneous breathing anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: non-intubation group: thoracic paravertebral nerve block was performed before anesthesia induction,after anesthesia induction laryngeal mask airway(LMA) is placed.
  intubation group:were given routine induction with double-lumen endotracheal intubation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spontaneous breathing anesthesia non-intubation group (Experimental): In this group all the patients with spontaneous breathing anesthesia
  Interventions: Procedure: General anesthesia with preservation of spontaneous breathing
- general anesthesia with double-lumen endotracheal intubation group (No Intervention): In this group all the patients with tradition anesthesia with double-lumen endotracheal intubation

INTERVENTIONS:
Procedure: General anesthesia with preservation of spontaneous breathing — non-intubation group, thoracic paravertebral nerve block was performed before anesthesia induction,when the BIS value drops to between 40 and 60, laryngeal mask airway(LMA) is placed,and observation of breathing
  Arms: spontaneous breathing anesthesia non-intubation group

SUMMARY:
the aim of this study is to evaluate the advantages of the non-intubation compared with intubation anesthesia on enhanced recovery after thoracoscopic surgery

DETAILED DESCRIPTION:
All patients will be screened to determine eligibility for study entry, and the patients who meet the eligibility requirements will be informed about the study and potential risks. After giving written informed consent, The patients were randomly divided into non-intubation group and intubation group

ELIGIBILITY:
Inclusion Criteria:

* age 18-69 years old
* Body mass index (BMI) was 18-24 kg / m2
* American Society of Anesthesiologists' physical classification class I-II
* The preoperative pulmonary function was normal

Exclusion Criteria:

* Severe cardiopulmonary disease
* Severe nervous system diseases
* Severe blood system diseases
* Severe liver and kidney dysfunction
* Conversion to thoracotomy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
the hospitalized stay | 1 year
  the hospitalized stay

SECONDARY OUTCOMES:
Visual analogue score (VAS) after operation; | 1 year
  Visual analogue score (VAS) was compared between the two groups
The postoperative complications | 1 year
  postoperative nausea and vomiting(PONV), pulmonary infection, atelectasis, sore throat, hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: sun caixia, doctor, Study Director — Department of Anesthesiology, Affiliated People's Hospital of Jiangsu University
Locations (1):
- Affiliated People's Hospital of Jiangsu University, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Data are available after publication and up to one year after publication
Access Criteria: Send an email to zhengyf.163@163.com

REFERENCES:
- [Background] Zheng H, Hu XF, Jiang GN, Ding JA, Zhu YM. Nonintubated-Awake Anesthesia for Uniportal Video-Assisted Thoracic Surgery Procedures. Thorac Surg Clin. 2017 Nov;27(4):399-406. doi: 10.1016/j.thorsurg.2017.06.008. PMID 28962712
- [Result] Hung WT, Cheng YJ, Chen JS. Video-Assisted Thoracoscopic Surgery Lobectomy for Lung Cancer in Nonintubated Anesthesia. Thorac Surg Clin. 2020 Feb;30(1):73-82. doi: 10.1016/j.thorsurg.2019.09.002. PMID 31761286
- [Result] AlGhamdi ZM, Lynhiavu L, Moon YK, Moon MH, Ahn S, Kim Y, Sung SW. Comparison of non-intubated versus intubated video-assisted thoracoscopic lobectomy for lung cancer. J Thorac Dis. 2018 Jul;10(7):4236-4243. doi: 10.21037/jtd.2018.06.163. PMID 30174869
- [Result] Kocaturk C, Kutluk AC, Usluer O, Onat S, Cinar HU, Yanik F, Cesur E, Ulku R, Karamustafaoglu A, Celik B, Demirhan R, Kalafat CE, Ozpolat B. Comparison of awake and intubated video-assisted thoracoscopic surgery in the diagnosis of pleural diseases: A prospective multicenter randomized trial. Turk Gogus Kalp Damar Cerrahisi Derg. 2019 Oct 23;27(4):550-556. doi: 10.5606/tgkdc.dergisi.2019.18214. eCollection 2019 Oct. PMID 32082924
- [Result] Senturk JC, Kristo G, Gold J, Bleday R, Whang E. The Development of Enhanced Recovery After Surgery Across Surgical Specialties. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):863-870. doi: 10.1089/lap.2017.0317. Epub 2017 Aug 10. PMID 28795911
- [Result] Guo Z, Shao W, Yin W, Chen H, Zhang X, Dong Q, Liang L, Wang W, Peng G, He J. Analysis of feasibility and safety of complete video-assisted thoracoscopic resection of anatomic pulmonary segments under non-intubated anesthesia. J Thorac Dis. 2014 Jan;6(1):37-44. doi: 10.3978/j.issn.2072-1439.2014.01.06. PMID 24455174
- [Result] Gonzalez M, Abdelnour-Berchtold E, Perentes JY, Doucet V, Zellweger M, Marcucci C, Ris HB, Krueger T, Gronchi F. An enhanced recovery after surgery program for video-assisted thoracoscopic surgery anatomical lung resections is cost-effective. J Thorac Dis. 2018 Oct;10(10):5879-5888. doi: 10.21037/jtd.2018.09.100. PMID 30505496
- [Result] Krediet AC, Moayeri N, van Geffen GJ, Bruhn J, Renes S, Bigeleisen PE, Groen GJ. Different Approaches to Ultrasound-guided Thoracic Paravertebral Block: An Illustrated Review. Anesthesiology. 2015 Aug;123(2):459-74. doi: 10.1097/ALN.0000000000000747. PMID 26083767
- [Result] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Result] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Result] Shen C, Che G. Tubeless minimally invasive treatment: taking a new step in enhanced recovery after surgery (ERAS). Thorac Cancer. 2019 Nov;10(11):2067-2070. doi: 10.1111/1759-7714.13206. Epub 2019 Oct 7. No abstract available. PMID 31588634
- [Result] Liu J, Cui F, Li S, Chen H, Shao W, Liang L, Yin W, Lin Y, He J. Nonintubated video-assisted thoracoscopic surgery under epidural anesthesia compared with conventional anesthetic option: a randomized control study. Surg Innov. 2015 Apr;22(2):123-30. doi: 10.1177/1553350614531662. Epub 2014 May 12. PMID 24821259
- [Result] Huang QW, Li JB, Huang Y, Zhang WQ, Lu ZW. A Comparison of Analgesia After a Thoracoscopic Lung Cancer Operation with a Sustained Epidural Block and a Sustained Paravertebral Block: A Randomized Controlled Study. Adv Ther. 2020 Sep;37(9):4000-4014. doi: 10.1007/s12325-020-01446-3. Epub 2020 Jul 31. PMID 32737760
- [Result] Chen N, Qiao Q, Chen R, Xu Q, Zhang Y, Tian Y. The effect of ultrasound-guided intercostal nerve block, single-injection erector spinae plane block and multiple-injection paravertebral block on postoperative analgesia in thoracoscopic surgery: A randomized, double-blinded, clinical trial. J Clin Anesth. 2020 Feb;59:106-111. doi: 10.1016/j.jclinane.2019.07.002. Epub 2019 Jul 19. PMID 31330457
- [Result] El-Boghdadly K, Madjdpour C, Chin KJ. Thoracic paravertebral blocks in abdominal surgery - a systematic review of randomized controlled trials. Br J Anaesth. 2016 Sep;117(3):297-308. doi: 10.1093/bja/aew269. PMID 27543524
- [Result] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Result] Janik M, Juhos P, Lucenic M, Tarabova K. Non-intubated Thoracoscopic Surgery-Pros and Cons. Front Surg. 2021 Dec 6;8:801718. doi: 10.3389/fsurg.2021.801718. eCollection 2021. PMID 34938770
- [Result] Qi L, Chen K, Luo B, Mao G, Pan L, Huang H, Li J, Chen S. Clinical application of preserving spontaneous breathing non-intubation anesthesia in thoracoscopic surgery for lung cancer under ERAS concept. Asia Pac J Clin Oncol. 2022 Oct;18(5):e329-e337. doi: 10.1111/ajco.13726. Epub 2021 Nov 24. PMID 34818467
- [Result] Cai LS, Hou B, Jin H, Bo Y, Chen XL, Dai J, Yang T, Lan BS, Ye J, Peng H, Peng J. Clinical evaluation of the rapid recovery of patients who underwent video-assisted thoracoscopic lung surgery under non-intubated anesthesia. Ann Transl Med. 2021 Dec;9(24):1783. doi: 10.21037/atm-21-6434. PMID 35071477